CLINICAL TRIAL: NCT02952235
Title: A Single Center, Randomized, Split-Face, Double-Blinded, Single Sun Exposure Evaluation of Sunscreens of SPF 50+ and Above Under Actual Use Conditions
Brief Title: Evaluation of Sunscreens Under Actual Use Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: CO-151112132858-SACT
Record Dates: First submitted 2016-10-31; First posted 2016-11-02 (Estimated); Last update posted 2017-06-08 (Actual); Status verified 2017-06

CONDITIONS: Sun Protection
MeSH Terms: interventions — Sunscreening Agents

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SPF50+ (Other): SPF 50+ assigned to Left side of face SPF 100+ assigned to Right side of face
  Interventions: Other: SPF50+
- SPF100+ (Other): SPF 100+ assigned to Left side of face SPF 50+ assigned to Right side of face
  Interventions: Other: SPF100+

INTERVENTIONS:
Other: SPF50+ — Sun protection
  Other Names: Sunscreens
  Arms: SPF50+
Other: SPF100+ — Sun protection
  Other Names: Sunscreens
  Arms: SPF100+

SUMMARY:
Use of two high SPF sunscreens under actual use conditions.

DETAILED DESCRIPTION:
To evaluate the difference in the level of sunburn (erythema) protection following a single period of natural sunlight exposure afforded by application of SPF 50+ and SPF 100+ sunscreens.

ELIGIBILITY:
Inclusion Criteria:

1. Males and Females with Fitzpatrick Skin Types I-III
2. At least 18 years old
3. Able to read, write, speak and understand the English language.
4. Has personally read, signed, and dated the Informed Consent Form (including HIPAA disclosure) and Photograph Release
5. Generally in good health based on medical history reported by the subject
6. Healthy male or female subjects with no history or evidence of clinically relevant medical disorder, as determined from a brief medical history interview.
7. Willing and able to follow the study instructions, including:

Remain outdoors for at least 5 hours on Day 1 during the study with face and neck uncovered (as much as possible)

* Apply the test products (sunscreen) to designated sides of the face and neck
* Remove any make-up, sunscreen, or other facial products at baseline prior to applying test product. Use test product in place of current sun protection topical skincare products (this includes make-up)
* Attend scheduled visits and intend to successfully complete the study
* Return ALL study products at Day 2 exit visit
* Refrain from using other sunscreen products or tanning bed use during the duration of the study.

Exclusion Criteria:

1. Individuals with known allergies or sensitivities to sunscreens or any ingredient contained in the test products or common topical skincare products, including adhesives.
2. Observable Sunburn (erythema score above 0.5) on the face and neck as determined by the PI or designee.
3. Women known to be pregnant or nursing.
4. Individuals with any disease or condition of the skin (e.g., active [i.e. flaring] eczema or psoriasis, skin cancer, polymorphic light eruption (PMLE), systemic lupus erythematous (SLE), xerodermapigmentosa) that could interfere with the study or increase risk to the subject.
5. Individuals with self-reported UNCONTROLLED metabolic conditions, such as diabetes, hypertension, hyper/hypothyroidism, hypercholesterolemia
6. Subjects who are taking medication for chronic conditions that may make a subject more sun sensitive (e.g., Tetracyclines, antifungals, certain diuretics, etc.)
7. Skin diseases on tested sites (e.g., photosensitivity disorders, etc.), which may influence the outcome of the study
8. Wearing of a full head covered ski mask.
9. An individual who has any condition which in the PI's judgment makes the candidate an inappropriate subject for study participation
10. Subjects who are related to those persons involved directly or indirectly with the conduct of this study (i.e., PI, sub-investigators, study coordinators, other site personnel, employees of Johnson & Johnson subsidiaries, contractors of Johnson & Johnson, and the families of each)
11. Individuals with a condition or situation which, in the PI's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study
12. Individual viewed by the PI as not being able to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Side-by-side Comparison (overall difference) of Sunburn. | Day 2
  The side-by-side comparison utilized the following condensed two side overall difference scale: L1 = subject's left side noticeably more sunburned than right side, 0= no difference in sunburn, R1= subject's right side noticeably more sunburned than left side. The 0 outcomes were excluded from the analysis.

SECONDARY OUTCOMES:
Difference in Erythema Score Between Left and Right Sides at Day 2 | Day 2
  Erythema was assessed using a scale of 0 = no burn, 1 = possible burn, not clearly defined; 2 = defined redness clearly caused by UV; 3 = severe sunburn with pronounced redness; and 4 = edema and blisters

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Williams, PhD, Study Director — Sponsor GmbH

IPD SHARING:
Plan to Share IPD: No